CLINICAL TRIAL: NCT04194073
Title: NightOwl SpO2 Calibration Study
Acronym: NOSCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ectosense NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19/0073/U
Record Dates: First submitted 2019-12-07; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Pulse Oximeter Calibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulse oximeter calibration population (Experimental): All subjects within this single arm of the study will undergo the calibration experiment as described in the Detailed Description
  Interventions: Device: Pulse oximeter calibration population (NightOwl)

INTERVENTIONS:
Device: Pulse oximeter calibration population (NightOwl) — The NightOwl is a finger and/or forehead mounted device with, among other functions, the capability to acquire double-wavelength PPG, from which SpO2 can be derived

SUMMARY:
Calibration of a software module that computes Oxygen saturation(SpO2) based on photoplethysmography (PPG) traces acquired by the NightOwl reflectance-based PPG sensor which is placed on the finger.

The study is designed in accordance with Medical electrical equipment - Part 2-61: Particular requirements for basic safety and essential performance of pulse oximeter equipment (ISO 80601- 2-61:2011)

DETAILED DESCRIPTION:
1. Trial objectives The main objective of this trial is to calibrate the parameters of a software module that computes SpO2 from the digitized raw red and infrared PPG traces of the NightOwl sensor placed at the fingertip. A CO-oximeter subsequently analyses the blood samples to derive "Gold-standard" SaO2 values to which the SpO2 samples can be compared. To obtain a spectrum of SpO2 levels between 100 and 73 % of healthy subjects, FiO2 will be progressively decreased in a hypoxia chamber under the guidance of an anaesthesiologist.
2. Endpoints Computation of Arms, the performance metric proposed by ISO 80601-2-61:2011 Annex CC: Determination of accuracy. This metric captures the bias and precision of the computed SpO2 values compared to the gold standard blood gas analysis method. The software modules' SpO2 computation accuracy (defined as Arms) will first be compared using the temporally paired oxygen saturation (SaO2) readings of the CO-oximeter benchmark.
3. Trial Design The trial is designed as open blind, non-randomized trial for clinical data acquisition. Approximately 10 healthy subjects will be included in the study.

Groups of up to 3 subjects will enter a hypoxia chamber. These subjects will have six NightOwl sensors attached, one placed on the index, middle, and ring finger of each hand. For each patient, one Nonin pulse oximeter with a real time SpO2 display will be placed on the pinkie, such that the SpO2 values can be monitored in real time. The NightOwl will transfer data to a smartphone, which serves as a data acquisition hub during the study. Once all sensors have been attached and data acquisition has started, FiO2 (percentage of oxygen in the space being measured) of the hypoxia chamber will gradually and be lowered over a course of approximately 2 hours, under the guidance of an anaesthesiologist. The investigators will attempt to create 5 stable plateaus of FiO2 values to allow for arterial blood sample drawing of a stable SaO2 value. As soon as SpO2 measured by a Nonin device of any subject drops below 73% for one minute, this particular subject will leave the hypoxia chamber immediately. As soon as all subjects have left the chamber, FiO2 will be returned to the oxygen level of the environment. The above is repeated for the next group of subjects until the warranted number of subjects is reached. During the procedure, for each subject, approximately 25 arterial blood samples will be drawn from an arterial catheter, of which the exact time of extraction will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with American Society of Anaesthesiologists health score (ASA) of 1 or 2, upon signing of informed consent.
* 15% of the study population or 2 subjects (whichever is larger) with dark pigmented skin should be included in the study

Exclusion Criteria:

* smokers or individuals exposed to high levels of carbon monoxide that result in elevated carboxyhemoglobin levels.
* individuals subject to conditions that result in elevated levels of methaemoglobin.

individuals with arterial cannulation or hypoxia at FiO2 = 0,21

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-12-07 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
A_rms determination | Within 3 months after subject recruitment, the calibration and A_rms determination should have been performed
  After calibration of the NightOwl SpO2 software module, the A_rms metric will be computed. This metric constitutes the performance metric proposed by ISO 80601-2-61:2011 Annex CC: Determination of accuracy. This metric captures the bias and precision of the computed SpO2 values compared to the benchmark.

CONTACTS AND LOCATIONS:
Overall Officials: Raf De Jongh, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- CMC, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No